CLINICAL TRIAL: NCT03828201
Title: Prospective, Randomized, Partially Blinded, Phase 2 Study of the Efficacy and Tolerability of Bedaquiline, Delamanid, Levofloxacin, Linezolid, and Clofazimine for Treatment of Patients With MDR-TB
Brief Title: Efficacy and Tolerability of Bedaquiline, Delamanid, Levofloxacin, Linezolid, and Clofazimine to Treat MDR-TB
Acronym: DRAMATIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Pfizer (Industry); Otsuka Pharmaceutical Co., Ltd. (Industry); University of California, San Francisco (Other); Westat (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Colorado, Denver (Other); Harvard Medical School (HMS and HSDM) (Other); National Lung Hospital, Vietnam (Unknown); De La Salle Health Sciences Institute, Philippines (Unknown)
Responsible Party: Principal Investigator, Charles R Horsburgh, Professor of Epidemiology, Boston University, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H39017; U01AI152980 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: bedaquiline (BDQ); delamanid (DLM); linezolid (LZD); levofloxacin (LFX); clofazimine (CF)
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — OPC-67683; Levofloxacin; bedaquiline; Clofazimine; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Investigational: DRAMATIC-16 weeks (Experimental): delamanid 300 mg orally, by mouth (PO) once a day (QD), 16 weeks levofloxacin 1000 mg PO QD, 16 weeks clofazimine 100 mg PO QD, 16 weeks bedaquiline 200 mg PO QD x 8 wk then 100 mg PO QD remainder linezolid 600 mg PO QD, Initial 16 weeks only
  Interventions: Drug: Delamanid; Drug: Levofloxacin; Drug: Bedaquiline; Drug: Clofazimine; Drug: Linezolid
- Investigational: DRAMATIC-24 weeks (Experimental): delamanid 300 mg orally, by mouth (PO) once a day (QD), 24 weeks levofloxacin 1000 mg PO QD, 24 weeks clofazimine 100 mg PO QD, 24 weeks bedaquiline 200 mg PO QD x 8 wk then 100 mg PO QD remainder linezolid 600 mg PO QD, Initial 16 weeks only
  Interventions: Drug: Delamanid; Drug: Levofloxacin; Drug: Bedaquiline; Drug: Clofazimine; Drug: Linezolid
- Investigational: DRAMATIC-32 weeks (Experimental): delamanid 300 mg orally, by mouth (PO) once a day (QD), 32 weeks levofloxacin 1000 mg PO QD, 32 weeks clofazimine 100 mg PO QD, 32 weeks bedaquiline 200 mg PO QD x 8 wk then 100 mg PO QD remainder linezolid 600 mg PO QD, Initial 16 weeks only
  Interventions: Drug: Delamanid; Drug: Levofloxacin; Drug: Bedaquiline; Drug: Clofazimine; Drug: Linezolid
- Investigational: DRAMATIC-40 weeks (Experimental): delamanid 300 mg orally, by mouth (PO) once a day (QD), 40 weeks levofloxacin 1000 mg PO QD, 40 weeks clofazimine 100 mg PO QD, 40 weeks bedaquiline 200 mg PO QD x 8 wk then 100 mg PO QD remainder linezolid 600 mg PO QD, Initial 16 weeks only
  Interventions: Drug: Delamanid; Drug: Levofloxacin; Drug: Bedaquiline; Drug: Clofazimine; Drug: Linezolid

INTERVENTIONS:
Drug: Delamanid — Frequency: daily Route of administration: oral
  Delamanid is a medication used to treat tuberculosis. Specifically it is used, along with other antituberculosis medications, for active multidrug-resistant tuberculosis. It is taken by mouth.
  Other Names: Deltyba
Drug: Levofloxacin — Frequency: daily Route of administration: oral
  Levofloxacin is an antibiotic used to treat a number of bacterial infections including acute bacterial sinusitis, pneumonia, urinary tract infections, chronic prostatitis, and some types of gastroenteritis. Along with other antibiotics it may be used to treat tuberculosis.
  Other Names: Levaquin
Drug: Bedaquiline — Frequency: daily Route of administration: oral
  Bedaquiline is indicated for use as part of an appropriate combination regimen for pulmonary multidrug-resistant tuberculosis (MDR-TB) in adult patients when an effective treatment regimen cannot otherwise be composed for reasons of resistance or tolerability.
  Other Names: Sirturo
Drug: Clofazimine — Frequency: daily Route of administration: oral
  Clofazimine has shown activity against multidrug-resistant tuberculosis (MDR-TB) and is now recommended by the World Health Organization (WHO) to treat drug resistant tuberculosis as a "Group B" drug. It is thought that clofazimine acts by inhibiting the formation of matrixes within the DNA and thus delaying the growth of the bacterium. Clofazimine first received FDA approval in 1986, although its use in the treatment of MDR-TB has not been approved by any stringent regulatory authorities and it is therefore used "off-label" for this function.
  Other Names: Lamprene
Drug: Linezolid — Frequency: daily Route of administration: oral
  Linezolid is an antibiotic used for the treatment of infections caused by Gram-positive bacteria that are resistant to other antibiotics.
  Other Names: Zyvox

SUMMARY:
Multidrug-resistant tuberculosis (MDR-TB) is tuberculosis (TB) that is resistant to at least isoniazid and rifampicin, the two most important anti-TB drugs. It occurs in 3.6% of newly diagnosed TB patients in the world and 17% of patients who have been previously treated. In 2017, approximately 600,000 people were estimated to have acquired MDR-TB. However, only 25% of persons with MDR-TB were diagnosed and started on treatment, reflecting inadequate diagnostic capacity and lack of TB treatment capacity.

In this multicenter, randomized, partially blinded, four-arm, phase 2 study, the investigators will examine the efficacy and safety of an all-oral regimen of bedaquiline, delamanid, levofloxacin, linezolid, and clofazimine given for 16, 24, 32 or 40 weeks

DETAILED DESCRIPTION:
Multidrug-resistant tuberculosis (MDR-TB) is tuberculosis that is resistant to at least isoniazid and rifampicin, the two most important drugs in treating TB. In 2017, approximately 558,000 new people were estimated to have developed MDR-TB, and 8.5% of the cases had extensively drug-resistant tuberculosis (XDR-TB).(1) Current WHO-endorsed MDR-TB treatment regimens take 9-20 months to complete and are associated with substantial toxicity, including deafness from injectable agents, hepatitis from pyrazinamide and severe neuropathy from linezolid. Given the long duration and toxicities of MDR-TB regimens, it is perhaps not surprising that WHO reports that only 25% of patients with MDR-TB are enrolled into WHO-endorsed treatment regimens. Thus, there is an urgent need for shorter, less toxic treatments for MDR-TB. This proposal will determine the efficacy, safety, tolerability and optimal duration of a novel, all oral MDR-TB treatment regimen while addressing three major challenges with innovations that have the potential to transform future trials.

The proposed DRAMATIC (Duration Randomized Anti-MDR-TB And Tailored Intervention Clinical) Trial is a multicenter, randomized, partially blinded, four-arm, phase 2 trial that will examine an injectable- and pyrazinamide-sparing regimen of bedaquiline, delamanid, levofloxacin, linezolid, and clofazimine. The DRAMATIC regimen limits the administration of linezolid to the initial 8 weeks of treatment, the window before linezolid-related neuropathy occurs. Animal and human studies provide evidence for the potential efficacy of this 5-drug regimen, but the optimal duration of treatment remains uncertain.(2-4)

Primary Objectives:

1. Describe the relationship between the duration of the experimental regimen and the proportion of participants with sustained cure at 76 weeks after randomization without treatment failure or relapse.
2. Describe the relationship between baseline prognostic risk strata and sustained cure at 76 weeks after randomization without treatment failure or relapse.
3. Evaluate the association between novel biologic markers and sustained cure at 76 weeks after randomization without treatment failure or relapse.

   Secondary Objectives:
4. Identify the shortest duration of the study regimen that has acceptable safety and efficacy for a Phase 3 clinical trial of the DRAMATIC regimen for treatment of MDR-TB.
5. Describe the frequency, magnitude, time course of and risk factors for QTc prolongation associated with the study regimen.
6. Demonstrate the feasibility and efficiency of implementing the new duration-randomized design in a multi-centre randomized trial of drug-resistant TB.
7. Determine if time to sputum culture conversion predicts optimal duration of treatment when stratified by extent of disease.
8. Describe the relationship between the duration of the experimental regimen and the proportion of participants with sustained cure at 104 weeks after randomization without treatment failure or relapse.
9. Assess vital status at 132 weeks post randomization.

Development of a shorter, better-tolerated treatment regimen will greatly enhance the ability of TB control programs to treat the growing number of patients. The DRAMATIC Trial will employ an innovative and efficient new design to establish a robust, nontoxic MDR-TB treatment regimen and identify the minimal duration for which it needs to be administered. These results will speed the process of moving forward to a confirmatory phase 3 clinical trial and increase the likelihood that such a trial is successful.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age ≥12 years. Prior to study procedures, if ≥18 years of age, provides informed consent; if <18 years of age, child provides informed assent and has a parent or guardian who provides informed consent on the participant's behalf.
2. Has pulmonary TB based on investigator assessment of all available information (e.g., chest radiograph, sputum smear, culture, molecular testing).
3. Has a sputum sample that is positive for M. tuberculosis that is rifamycin-resistant and fluoroquinolone-susceptible by molecular assay.
4. Is HIV seropositive or seronegative; HIV serostatus must be assessed at screening if either (a) HIV serostatus is unknown, or (b) the last documented negative HIV test was more than two (2) months prior to screening.
5. Willing to attend scheduled follow-up visits and undergo study assessments.
6. Participants of child-bearing potential must agree either (a) to practice an adequate birth control (defined as one of the following oral contraceptives, intrauterine devices, contraceptive implants under the skin, contraceptive rings or patches or injections, diaphragms with spermicide or condoms with foam) or (b) to abstain from heterosexual intercourse during study regimen.

Exclusion Criteria:

1. Current MTB isolate is known at screening to be fluoroquinolone-resistant.
2. History of allergy (hypersensitivity) or intolerability to one or more agents in the investigational regimens (i.e., Arms 1 and 2)
3. History of serotonin syndrome
4. History of symptomatic ventricular arrhythmia or is taking anti-arrhythmic agents
5. History of optic neuropathy or peripheral neuropathy
6. History of Ehlers-Danlos Syndrome, Marfan Syndrome or aortic aneurism
7. History of prior treatment with delamanid or linezolid for TB for greater than one month.
8. Has at screening received ≥14 days of second-line anti-TB drugs during current TB episode
9. Has at screening a Karnofsky score of ≤40 or, in the opinion of the Investigator, is unlikely to survive 76 weeks.
10. Has at screening laboratory results that meet one or more of the following criteria:

    * Hemoglobin concentration 8.0 g/dL (<80 g/L)
    * Platelet count of <80,000/mm3
    * Absolute neutrophil count (ANC) <2000/ mm3
    * Serum creatinine >2.0 mg/dL (>177 µmol/L)
    * Serum ALT >3x upper limit of normal (ULN)
    * Total bilirubin >3x upper limit of normal (ULN)
    * Serum albumin <2.8 g/dL (<28 g/L)
    * For women of childbearing potential, a positive or indeterminate serum pregnancy test
11. For women of childbearing potential, has a positive or indeterminate urine pregnancy test on the day of randomization.
12. Has at screening a mean QTcF >450 msec based on three ECGs.
13. At screening requires ongoing use of prohibited drugs indicated in section 4.2
14. At screening, has weight less than 33 Kg
15. In the investigator's judgement is unable to provide consent (if ≥18 years of age) or unable to provide assent (if >12 years of age).
16. History of congestive heart failure

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Efficacy - Frequency of "successful treatment" outcomes | Week 76
  A participant's outcome will be classified as successful if, at 76 weeks after initiation of treatment, they have a "negative" sputum culture and were not previously classified as unsuccessful; if the participant is unable to produce sputum at that time, the outcome will be classified as successful if they had a negative culture result at the last visit at which they had a sputum culture result.
  A participant's outcome will be classified as unsuccessful if any of the following occur prior to week 76: Addition or replacement of 2 or more anti-tuberculosis (TB) drugs from the assigned regimen, the participant has a positive culture for M. tuberculosis and that isolate is not demonstrated to be genetically different from the initial isolate, undergoing surgery for multidrug-resistant TB (MDR-TB), lost to follow-up, surgery for MDR-TB, extended treatment, and death.
Treatment Safety - Frequency of participants with grade 3, 4, or 5 adverse events | 44 weeks
  The primary outcome for safety are Grade 3, 4, or 5 adverse events

SECONDARY OUTCOMES:
Efficacy outcome- Frequency of participants who survive | Week 132
  Evaluate survival at 132 weeks post randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Horsburgh, MD, Principal Investigator — Boston University; Payam Nahid, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- De La Salle Health Sciences Institute, Dasmariñas, Philippines
- National Lung Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No